CLINICAL TRIAL: NCT00128063
Title: A Phase 1 & 2, Randomized Open-Label Study to Evaluate the Pharmacokinetics, Safety and Antiretroviral Activity of Succinylated Human Serum Albumin (Suc-HSA) in Treatment Naïve HIV-1 Infected Subjects
Brief Title: Succinylated Human Serum Albumin (Suc-HSA) for HIV-1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Antiviral Therapy Evaluation Center (Other)
Collaborators: University Medical Center Groningen (Other); Prothya Biosolutions (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-IAT-0047
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infections
Keywords: HIV-1; succinylated human serum albumin; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: succinylated human serum albumin

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetic behavior of Suc-HSA after consecutive daily intravenous (i.v.) doses. The secondary objectives are to evaluate the safety and tolerability and the antiretroviral and immunological effects of consecutive daily i.v. doses of Suc-HSA.

DETAILED DESCRIPTION:
This is a single centre, single arm study. Subjects will receive 5 consecutive daily doses of Suc-HSA at a dose of 10 mg/kg on days 0, 1, 2, 3 and 4 on the Special Investigation Unit (SIU), with a safety follow up on the SIU for 4 hours on day 1 and 2 hours on the next days. There will be follow-up visits on week 1, 2, 4 and 12. Standard safety parameters (physical examination, clinical symptoms, laboratory hematology and biochemistry) will be followed until week 12. Plasma HIV-1 RNA and CD4+/CD8+ cell counts will be assessed at every visit. Plasma drug levels (trough and peak) will be measured from baseline until week 2.

6 patients will be included in this study as described in this protocol amendment.

Eligible subjects are chronic HIV-1 infected patients who have never been treated with antiretroviral treatment and for whom there is no need to start antiretroviral treatment.

Test Product: Suc-HSA, a candidate HIV-1 fusion inhibitor.

Duration of treatment: 5 days

Criteria for evaluation:

* Safety: symptoms, signs at physical examination, standard hematology and chemistry laboratory parameters- Efficacy: changes in plasma HIV-1 RNA and CD4+ T cell count
* Pharmacokinetics: plasma levels of Suc-HSA: Cmin, Cmax and AUC

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age;
2. Voluntarily signed informed consent;
3. Patient has a proven HIV-1 infection (with positive antibodies against HIV-1 and a detectable plasma HIV-1 RNA);
4. Patient is HIV-1 treatment naïve;
5. CD4+ T-cell count ≥ 350 x 10^6/L;
6. Plasma HIV-1 RNA level at screening visit of at least 5.000 copies/ml, and not varying more than ± 0.5 log10 copies during the preceding 6 month period;
7. Patient was participant in part 1 of the original Suc-HSA study (protocol no. 2003-002, version 2.4, dated 18 November 2003) and the administration of Suc-HSA occurred more than 8 weeks ago, OR patient was not participant in this study;
8. Patient is one of the following:

   * not heterosexually active, OR
   * a heterosexually active female, agreeing to use an effective method of contraception with her partner (combined oral contraceptive pill; injectable contraceptive; intrauterine contraceptive device (IUCD); consistent use of condoms if using these; physiological or anatomical sterility in herself or her partner) from 14 days prior to the first administration of study medication until 4 months after the last, and willing to undergo urine pregnancy tests prior to the first and last administration, OR
   * a heterosexually active male, agreeing to use an effective method of contraception with his partner from the day of the first administration until 4 months after the last administration.

Exclusion Criteria:

1. History of an AIDS defining event;
2. Use of antiretroviral or immunomodulatory therapy;
3. Any reason to start antiretroviral therapy at the time of enrolment or which is expected to occur during the course of the study at the time of enrolment;
4. Presence of active, replicating hepatitis B and/or C virus co-infection;
5. ASAT and/or ALAT > 3 times upper limit of normal (ULN) (AIDS Clinical Trials Group [ACTG] toxicity scale);
6. Serum creatinine measuring > 1.5 x ULN;
7. Total bilirubin > 2x ULN;
8. Neutropenia (absolute neutrophil count < 1000/mm3);
9. Presence of any clinically significant disease or findings during screening, that in the opinion of the investigator could compromise the safety of the subject;
10. Patient is female and (willing to become) pregnant or breast-feeding;
11. Any other condition which, in the opinion of the investigator, may interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic behavior of Suc-HSA after consecutive daily i.v. doses.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability and the antiretroviral and immunological effects of consecutive daily i.v. doses of Suc-HSA.

CONTACTS AND LOCATIONS:
Overall Officials: Joep MA Lange, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Jan Prins, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, University of Amsterdam, Amsterdam, North Holland, Netherlands